CLINICAL TRIAL: NCT06014463
Title: Evaluation of Adult Patients With Immunodeficiency Within the Scope of the International Classification of Functionality, Ability and Health
Brief Title: Evaluation of Adult Patients With Immunodeficiency Within the Scope of the ICF
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Baskent University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Associate Professor, Hacettepe University
Other Study IDs: GO 23/16
Record Dates: First submitted 2023-08-18; First posted 2023-08-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Primary Immune Deficiency; Exercise Capacity; Physical Activity; Quality of Life
Keywords: Primary Immune Deficiency; ICF; Functional Performance
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Primary Immune Deficiency: Patients between the ages of 18-65 years who have been diagnosed with primary immunodeficiency
- Healthy Controls: Age and sex matched healthy controls between the ages of 18-65 years

SUMMARY:
Primary immunodeficiency is a clinically, immunologically, and genetically heterogeneous group of diseases that occur as a result of quantitative and/or qualitative deficiency of one or more cellular and molecular components belonging to the immune system. This classification, called the International Classification of Functioning, Disability and Health ( ICF), constitutes a common language and perspective for the definition of health and health-related conditions. This study aimed to evaluate the body structure function, activity and participation limitations of adult immunodeficiency patients within the scope of ICF and to compare body structure function, activity and participation limitations and compare with healthy people.

DETAILED DESCRIPTION:
Primary immunodeficiency is a clinically, immunologically and genetically heterogeneous group of diseases that occur as a result of quantitative and/or qualitative deficiency of one or more cellular and molecular components belonging to the immune system. The overall prevalence of PID in the world is stated as 1/2,000-1/10,000 per live birth. In our country, the national PID registration system has just been established. It is estimated that this rate is higher in developing countries such as Turkey, where there is a lot of inbreeding. The clinical appearance of PID is highly variable; however, most often it is characterized by an increased predisposition to infection. Therefore, the disease manifests itself with infections that are "recurrent and difficult to respond to treatment". PID, which mostly starts to give symptoms in childhood, are in the category of rare diseases. For this reason, the probability of receiving a diagnosis in primary and second-line healthcare institutions is very low. Since the course of the disease is poor in a significant part of PID, early diagnosis and timely treatment are very important for reducing mortality, morbidity and economic burden. This is possible with the level of social awareness and the high index of suspicion of medical personnel. For the successful management of the disease, the patient should be quickly referred to a clinical immunologist experienced in immunodeficiencies and further tests should be performed. Fifteen years ago, the Jeffrey Modell Foundation (JMF) identified clinical signs that arouse suspicion of PID in children and adults. This document is a useful basis, but revision is required because it does not take into account the autoimmune, inflammatory or malignant manifestations of PID, which may be the cause of the main clinical presentation in some of the PID. Pulmonary complications are common in PID and contribute significantly to the morbidity and mortality of patients. Recurrent respiratory infections (more than 2 per year for children and within 3 years for adults) are one of the 10 warning signs of PİY recommended by the Jeffrey Modell Foundation and are often the cause of death in adults with PID. Especially in PID, which is characterized by antibody deficiency, frequent recurrent upper and lower respiratory tract infections lead to chronic complications in tissues and organs. Bronchiectasis is the prominent one among these. According to the European Society of Immunodeficiencies, bronchiectasis develops in ~23% of patients with NDI (one-third of all PID patients) . It has been shown that the general state of health, psychosocial well-being level and quality of life are low in patients with PI who have developed chronic lung disease, and it has been found that their daily activities are significantly limited.

This classification, called the International Classification of Functioning, Disability and Health (ICF), was developed in 2000 to create a common language and perspective for the definition of health and health-related conditions. Objectives of the ICF classification:

* To create a scientifically based approach to determine health and health-related conditions
* To facilitate and increase communication between all health professionals and individuals in different professional groups and to ensure the formation of a common language Dec
* To ensure the determination of health-related applications
* Coding health-related factors with a specific system ICF provides the functional status of individuals and the identification of problems that they may encounter in daily life from a biopsychosocial point of view.

ICF-CY evaluates health-related situations with a total of 1685 items in 4 sections. The fact that it has so much substance constitutes a disadvantage in terms of its use. For this reason, with the ICF Core Sets Project study in 2003, disease-specific core sets were created by selecting categories that are specific to diseases and can fully identify the patient. Core sets, just like ICF, treat the patient holistically. Each set has 2 separate forms in the form of short form and long form. There are 5 core sets that can evaluate cardiopulmonary system disorders. Cardiopulmonary disorders, obesity, diabetes mellitus, COPD, chronic ischemic heart problems are the core sets. In a study conducted on 40 pediatric patients with and without cystic fibrosis, it was shown that the ICF model is applicable and useful in evaluating body function and structure disorders such as November muscle weakness, postural anomalies, and limitations in activity and participation in daily life, and in creating a treatment plan. a study conducted on 24 lung transplant patients showed that the ICF model is practical and applicable in the clinic for evaluating activity and participation restrictions such as decreased exercise capacity, body structure and function disorders such as postural disorders, physical activity in daily life, balance disorder, decreased quality of life.

However, there are no studies evaluating the body structure, function, activity and participation of immunodeficiency patients within the scope of ICF. Our study has the feature of being the first study in which immunodeficiency patients were evaluated within the scope of ICF. With this study, the investigators believe that a holistic assessment conducted within the framework of ICF in immunodeficiency patients will have a positive impact on the clinical decision-making process of cardiopulmonary rehabilitation professionals. This study aims; to evaluate the body structure function, activity and participation limitations of adult immunodeficiency patients within the scope of ICF and to compare with healthy people. A second goal is to evaluate the relationships between body structure, function, activity and participation limitations in adult immune deficiency patients.

ELIGIBILITY:
Criteria for Inclusion in the Adult Immunodeficiency Group

1. to be between the ages of 18-65 years old.
2. to be volunteer to participate in research
3. to have been diagnosed with Primary Immunodeficiency
4. to be taking immunoglobulin replacement therapy
5. to have no problems in reading and/or understanding scales and being able to cooperate with tests

Criteria for exclusion of the Adult Immunodeficiency Group:

1. The presence of active infection
2. Musculoskeletal and neurological disease that may affect exercise performance symptomatic heart disease
3. To have a neurological disease or other clinical diagnosis that may affect cognitive status

Criteria for inclusion in the control group:

1. to be between the ages of 18-65 years old
2. to give informed consent
3. to have no problems in reading and/or understanding scales and being able to cooperate with tests

Criteria for exclusion of the Control Group:

1. to have any orthopedic or neuromuscular disorder that will interfere with walking or exercise performance,
2. to have any chronic disease or to have psychiatric disorders or mental influences that may prevent cooperation or compliance with exercise tests.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65 who have been diagnosed with immunodeficiency at Başkent University Hospital Immunology Department and Gülhane Hospital Immunology Department and who are willing to participate in the research and 18-65 patients who are diagnosed with immunodeficiency will be accepted for the study.
  The snowball sampling method will be used for our control group. We plan to contact the patient's relatives and then contact someone else in the same way. At the same time, we plan to prepare a text explaining each method and reach people through social media.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of hand grip strength | 1 day
  The participants will be measured in an unsupported sitting position with his back upright, while the elbow is in flexion (the person's arm is adjacent to the torso, in a neutral position, and the elbow is in a 90° flexion, with the wrist neutral). The measurements for the dominant and non-dominant sides will be repeated three times. The average of the three measurements for each side will be taken and recorded in Newton (N).

SECONDARY OUTCOMES:
Evaluation of body composition: | 1 day
  The bioelectric impedance analysis (XIAOMI MI 2 Body Analysis Scale)
Comorbidity Assessment | 1 day
  The Charlson Comorbidity Index developed by Charlson et al. will be used to determine the short-term mortality risk of patients with concomitant disease conditions. DM 1 point without myocardial infarction, congestive heart failure, peripheral vascular disease, cerebrovascular disease, dementia, chronic pulmonary disease, connective tissue disorder, peptic ulcer disease, mild liver disease and end-organ damage on the scale; hemiplegia, moderate and severe kidney disease, DM with end-organ damage, non-metastatic tumor, leukemia, lymphoma and myeloma are 2 points; 3 points for moderate or severe liver disease; and metastatic solid tumor or Acquired Immune Deficiency Syndrome (Acquired Immune Deficiency Syndrome -AIDS) is 6 points. The total score, on the other hand, will be calculated by adding up the equivalent scores of diseases.
Evaluation of Sleep Quality | 1 day
  The Pittsburgh Sleep Quality Index (PSQI), which has Turkish validity and reliability and evaluates an individual's sleep quality for the last one month, contains a total of 24 questions. 19 Of these questions are answered by the patient himself, he participates in the scoring. 5 questions are answered by the patient's spouse or roommate and are used only for clinical information and do not participate in scoring. Each question is evaluated with a score between 0-3.Dec. The total PSQI score takes a value between 0-21.Dec. In the end, 7 components are calculated. These; subjective sleep quality is sleep latency, sleep duration, habitual sleep efficiency, sleep disorder, sleeping medication use, daytime dysfunction. The total PSQI score is obtained by summing the scores of all these components. Those with a total score of 5 and below 5 are rated as having "good" sleep quality, and those with a total score of over 5 are rated as "poor" sleep quality.
Fatigue Assessment | 1 day
  The severity of fatigue in the daily life of the patients was evaluated with the Fatigue Severity Scale (FSS), which has validity and reliability in Turkish. Patients can apply this scale, which has nine items, on their own. The patient is informed about how to fill out the scale, but patients are not guided for questions and statements that they have difficulty understanding. Patients are asked to choose a score from 1 to 7, which indicates how much they agree with each statement on the scale. Statements related to scoring; 1. I Strongly Disagree, 2. Disagree, 3. I Tend to Disagree, 4: I am Undecided, 5: I Tend to Agree, 6: I Agree, 7: I Strongly Agree. Scores of 4 and above given to the statements indicate that fatigue is severe.
Posture Evaluation | 1 day
  The posture analysis form developed by Corbin and his colleagues was used to determine the postural disorders of the patients. The analysis will be evaluated in two different ways, posterior and lateral. According to the scoring of the results of the posture analyses according to their severity, they will be rated as 0: none, 1: light, 2: moderate and 3: severe. According to the total lateral and posterior posture score, the total score varies between 0-12. Dec.
Evaluation of Quality of Life | 1 day
  To evaluate the quality of life, Koçyiğit et al. the SF-36 quality of life scale, which has been validated by our country, will be applied. SF-36 Quality of Life consists of eight subgroups: physical function, physical role restriction, emotional role restriction, body pain, social function, mental health, vitality, general health and contains a total of 36 questions. Scoring is made between 0-100 for each group. The lowest score indicates the worst state of health. The last four weeks of the patients' conditions will be taken into account in the evaluation.
Evaluation of Daily Living Activities | 1 day
  To evaluate daily living activities, Işık et al. The Lawton Instrumental Daily Living Activities (IADL) scale, which has been made a validity study for our country, will be applied. The Lawton Instrumental Daily Living Activities (IADL) scale consists of eight categories: the ability to use a phone, shopping, food preparation, household chores, laundry, transportation method, responsibility for using one's medicines and the ability to manage financial affairs. The responses given to each of the eight categories on the scale are coded as 0 (can't or partially can) or 1 (can), and the responses are summed. The total score varies between 0 (low-functioning, dependent) and 8 December (high-functioning, independent).
Evaluation of Physical Activity | 7 day
  The International Physical Activity Questionnaire (IPAQ) long form, which has validity and reliability in Turkish, will be used to determine the level of physical activity by questioning the activities within the last 7 days. It includes the sum of the duration (how many minutes per day) and frequency (how many days in the last 7 days) to calculate the total score. The total score can be calculated with two different evaluations. The first includes special scoring (work, transportation, home gardening, leisure time), and the second includes activity-specific scoring (walking, moderate-intensity activity, vigorous activity). In activity-specific scoring, walking, moderate violent activity and violent activity under their heading of the sections are Decoupled by the sum between them. With these calculations, a value is found in MET-minutes. A MET-minute is calculated by multiplying the MET score by the minute of the activity performed.
Exercise Capacity Assessment | 1 day
  It is a simple, applicable alternative test to 6 DYT that evaluates exercise capacity, whose reliability has been proven in various lung diseases such as Cystic Fibrosis and COPD. The patient, whose height is 44 cm, who is sitting in a chair without armbands and has a place to recline, is asked to cross his arms to chest level. The patient, who is standing upright with his hips and knees coming to full flexion, sits down again. the number of repetitions of the patient who does sit-up for 1 minute will be recorded. In the interpretation of the test, the reference values determined by age will be taken as a basis and expressed as a percentage of the expected values. In addition, heart rate, oxygen saturation, dyspnea and leg fatigue values will be recorded before and after the test.
Evaluation of ICF Parameters | 1 day
  ICF belongs to the international classification "family" developed by the World Health Organization (WHO) for application in many areas of health. It uses a standard, common language that enables worldwide communication related to health and medical care in various disciplines and scientific fields. In order to evaluate disorders, activity limitations and limitations in participation, the subparagraphs of area b (body functions), area s (body structures), area d (activity and participation level) and area e (environmental and personal factors) will be comprehensively scanned to select items related to the classification area. Scoring is done separately for each item in the body structures (s), body functions (b), activity and participation (d), environmental and personal factors section. In this study, a Decrement between 0-4 will be made for each item in all sections. Items or sections with a higher score indicate more affect/disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik-Kutukcu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Ebru Çalık Kutukcu, Ankara, Hacettepe Unıversity, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No